CLINICAL TRIAL: NCT05488574
Title: Effects of Novel Breathing, Behavior Modification, Yoga Positioning Integrated Program on Weight Loss.
Brief Title: Effects of Novel Breathing Behavior Modification Yoga Positioning Integrated Program on Weight Loss
Acronym: Breathing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Touro University Nevada (Other)
Responsible Party: Principal Investigator, Michael Laymon, Professor, Director Human Performance Laboratory, Touro University Nevada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ML-CHHS-22-338
Record Dates: First submitted 2022-07-28; First posted 2022-08-04 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Weight Loss; Metabolism
Keywords: metabolism; obesity; mentation
MeSH Terms: conditions — Weight Loss; Obesity

STUDY DESIGN:
Intervention Model Description: A randomized control group, investigator blinded, repeated measure interventional program.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators doing data collection will not know which subjects are interventional and which are controls. Outcomes assessor will not be aware of which group of subjects were interventional and which did not participate in intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep breathing with Yoga positioning (Experimental): subjects participating in breathing and moving meditation program. 12 minutes daily of deep breathing and yoga positioning first 30 days, then continuation of breathing and positioning and self-directed, mentored, behavior modification activities the second 30 days.
  Interventions: Other: Deep breathing with Yoga positioning
- Control (No Intervention): No changes in lifestyle or activities over the 60 day period.

INTERVENTIONS:
Other: Deep breathing with Yoga positioning — Deep breathing with yoga positioning 10min in morning, 1 minute noon, and 1 minute evening (diner)
  Other Names: Novel breathing and mindfulness moving-meditation.
  Arms: Deep breathing with Yoga positioning

SUMMARY:
This study is to evaluate the physical and cognitive effects of a 15 min per day novel breathing and mindfulness moving-meditation program on metabolism, cognition, and emotion health. It is thought that the breathing and movement program will increase basal metabolism, facilitate fat loss, and decrease depressive behaviors. Anthropometric, blood chemistries, and cognitive measures of depression, sleep, and hunger will be measured over a two-month interventional program.

DETAILED DESCRIPTION:
Subjects will be randomized into two groups, an active group and control group. For the first 30 days, the active group will follow the movement/breath program and the controls will be instructed not to change their lifestyle (no change in diet, and no change in exercise / physical activities). The technicians taking measurements will be blinded as to which participants are actives vs controls. The following 30 days' intervention will consist of continuing the Phase I interventions combined with implementing the behavior change strategies on 2 to 3 habit changes self-selected from a list of 30 top "bad habits" that contribute to weight gain and undermine one's ability to lose weight with the control group again not changing any lifestyle activities. Measurements: Measurements will be taken at the start (baseline), 10 days, 30 days, and 60 days of intervention with the measurement days scheduled to evaluate people completing 10 full days of the program, 30 full days, and 60 full days respectively. Measurements taken at each interval to include weight, body composition (lean mass & fat percentages), anthropometric measurements (umbilicus, hips, right thigh, right upper arm), pO2, resting heart rate, HRV, blood pressure, pulmonary health (i.e., O2 max, spirometry), hunger, sleep, and depression rating (by self-assessment survey scale). Serum chemistry for basic metabolic panel, inflammatory markers, and lipids, hematology for oxygen carrying capacity and gross immune response, Human Growth Factor production via ELISA quantification, imaging ultrasound to measure subcutaneous fat thickness at the areas of girth measurements, DEXA for overall and targeted areas body composition, and resting metabolic rate via oxygen plethysmograph.

ELIGIBILITY:
Inclusion Criteria

* Age 18-70 years
* Body Mass Index at or above 27
* Stable weight past 3 months
* able to stand for 10 minutes
* Able to lift arms overhead

Exclusion Criteria:

* Chronic Obstructive Pulmonary Disease
* acute respiratory distress
* supplemental oxygen use
* inability to stand, flex trunk, or move arms overhead
* Pacemaker implant
* Taking beta blocking medications.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2022-11-23 (Estimated); Study Completion 2022-11-23 (Estimated)

PRIMARY OUTCOMES:
Change rom baseline in body Weight | Baseline, 10 days, 30 days, and 60 days.
  Weight in kilograms
Change from baseline in Body Mass Index | Baseline, 10 days, 30 days, and 60 days.
  DEXA Measurement of % total fat

SECONDARY OUTCOMES:
Human Growth Hormone - Metabolic rate | baseline, 10 days, 30 days, 60 days
  Measurement of Human Growth Hormone
VO2 at rest, Oxygen consumption at rest-resting metabolic rate(RMR) | Baseline, 10 days, 30 days, and 60 days.
  Oxygen consumption via oxygen plethysmograph
Respiratory quotient (RQ) - metabolic rate | Baseline, 10 days, 30 days, and 60 days.
  CO2 eliminated/O2 consumed
lipid panel - metabolic rate | Baseline, 10 days, 30 days, and 60 days.
  Total cholesterol, high density lipids, low density lipids, triglycerides

OTHER OUTCOMES:
stress level - autonomic function | Baseline, 10 days, 30 days, 60 days
  Heart Rate Variability
Depression | Baseline, 10 days, 30 days, and 60 days.
  Hamilton Depression Rating Scale (HAM-D) depression index self reported survey scored 0-62 with higher score indicating a worse outcome.
Sleep | Baseline, 10 days, 30 days, and 60 days.
  Insomnia Severity Index (ISI) self reported survey scored 0-28 with higher score indicating worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Laymon, DSc, PT, Principal Investigator — Touro University Nevada
Locations (1):
- Michael Laymon, Henderson, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
To protect privacy of subjects, Data will be reported as cumulative without individual participant data. In the event of potential health adverse disease process IPD may be shared with individuals' consent to their designated, licensed, healthcare provider.

REFERENCES:
- [Result] Sato K, Kawamura T, Yamagiwa S. The "Senobi" breathing exercise ameliorates depression in obese women through up-regulation of sympathetic nerve activity and hormone secretion. Biomed Res. 2011 Apr;32(2):175-80. doi: 10.2220/biomedres.32.175. PMID 21551954
- [Result] Sato K, Kawamura T, Yamagiwa S. The "Senobi" breathing exercise is recommended as first line treatment for obesity. Biomed Res. 2010 Aug;31(4):259-62. doi: 10.2220/biomedres.31.259. PMID 20834183
- [Result] Sato K, Kawamura T, Abo T. "Senobi" stretch ameliorates asthma symptoms by restoring autonomic nervous system balance. J Investig Med. 2010 Dec;58(8):968-70. doi: 10.231/JIM.0b013e3181f9167b. PMID 20930645
- [Result] Nivethitha L, Mooventhan A, Manjunath NK. Evaluation of Cardiovascular Functions during the Practice of Different Types of Yogic Breathing Techniques. Int J Yoga. 2021 May-Aug;14(2):158-162. doi: 10.4103/ijoy.IJOY_61_20. Epub 2021 May 10. PMID 34188389
- [Result] Nivethitha L, Mooventhan A, Manjunath NK, Bathala L, Sharma VK. Cerebrovascular Hemodynamics During the Practice of Bhramari Pranayama, Kapalbhati and Bahir-Kumbhaka: An Exploratory Study. Appl Psychophysiol Biofeedback. 2018 Mar;43(1):87-92. doi: 10.1007/s10484-017-9387-8. PMID 29188396